CLINICAL TRIAL: NCT00127543
Title: Kid Cards: Teaching Kids About Medicines
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not completed
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 05 06-089E
Record Dates: First submitted 2005-08-05; First posted 2005-08-08 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Hemophilia; Sickle Cell Disease; Neoplasms; Blood Coagulation Disorders
Keywords: Medication Education; Pediatric
MeSH Terms: conditions — Hemophilia A; Anemia, Sickle Cell; Neoplasms; Blood Coagulation Disorders

INTERVENTIONS:
Behavioral: Medication Education for Children

SUMMARY:
This study is being done to see if education about medicines directed toward children will improve their knowledge. The investigators also want to know if this knowledge lasts over time. Right now there are few medication instructional cards that are appropriate for children. Most of the medication cards provide information for adults. Some studies have shown that by teaching children directly, the children may take medicine at the right time for the right reason, have fewer side effects and know more about their medicine.

The purpose of this research study is to see if education about medication helps children learn more about their medicine and if this knowledge lasts.

DETAILED DESCRIPTION:
In 2004, then Surgeon General Carmona stated that a health literate individual is more apt to know the answer, when asked how to keep themselves well (AHRQ, 2004). There is a burgeoning movement among medical professionals to address health literacy. Teaching health information to children will empower them to actively participate in their current care and provide self-management skills that will assist them to keep themselves well throughout their lives. Currently, few medication administration instructional cards exist that are appropriate for children. Providing medication information that the child might understand may result in better administration compliance, fewer adverse effects and develop an individual that is knowledgeable regarding medications and appropriate administration. The purpose if this research is to develop medication administration cards, appropriate for children, which provide information on the most commonly used drugs among the Hematology/Oncology population.

The overall objective of this research is to develop medication informational cards for medications frequently used within the Hematology/Oncology pediatric population, and evaluate the effectiveness of these cards, by means of a pre- and post-test.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 7 - 11 years
* Currently receiving disease management primarily coordinated through the Hematology/Oncology section
* Receiving a medication identified as a variable for this study
* Are able to assent and have a parent/guardian who is willing to consent to study participation
* Suffer no apparent developmental difficulty that would prevent or make study participation difficult

Exclusion Criteria:

* Individuals who cannot read or write English
* Individuals who are known to be non-compliant with medication routine and/or adhering to follow-up visits.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-08; Study Completion 2006-04

PRIMARY OUTCOMES:
Develop medication cards appropriate for children
Develop a post-test to determine the effectiveness
Obtain data to support teaching children about medication

SECONDARY OUTCOMES:
Assess the clinical implications of this research

CONTACTS AND LOCATIONS:
Overall Officials: Heather E Curry, RN, MSN, Principal Investigator — Childrens Mercy Hospitals and Clinics
Locations (1):
- Childrens Mercy Hospitals and Clinics, Kansas City, Missouri, United States